CLINICAL TRIAL: NCT05879991
Title: A Phase I, Open-label Trial in Two Parallel Parts to Investigate Mass Balance, Metabolism, and Basic Pharmacokinetics of BI 1810631 (C-14) Administered as Oral Solution (Part A) and to Investigate Absolute Bioavailability of BI 1810631 Administered as Film-coated Tablet Together With an Intravenous Microtracer Dose of BI 1810631 (C-14) (Part B) in Healthy Male Volunteers
Brief Title: A Study in Healthy Men to Test How Zongertinib (BI 1810631) is Taken up and Processed by the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1479-0006; 2022-503047-17-00 (Registry Identifier: CTIS); U1111-1291-2883 (Registry Identifier: WHO registry)
Record Dates: First submitted 2023-05-25; First posted 2023-05-30 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Healthy
MeSH Terms: interventions — Carbon-14

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A - zongertinib (C-14) (T1) (Experimental): Healthy male subjects were administered a single oral dose of radioactively-labelled zongertinib (C-14) as a solution (test treatment 1 [T1]) with 240 milliliter (mL) of water, after an overnight fast of at least 10 hours (h).
  The solution contained a mixture of pure [14C]-labelled zongertinib ("hot") drug substance, and zongertinib, i.e. unlabeled ("cold") drug substance, and it contained a radioactive dose of approximately 3.7 Megabecquerel (MBq).
  Interventions: Drug: zongertinib (C-14)
- Part B - zongertinib (T2), then zongertinib (C-14) (R) (Experimental): Healthy male subjects were administered one zongertinib film-coated tablet (test treatment 2 [T2]) orally with 240 mL of water after an overnight fast of at least 10 h.
  Two hours later, subjects were administered a single solution of radioactively-labelled zongertinib (C-14) (reference treatment [R]) via intravenous infusion. The solution contained a mixture of pure [14C]-labelled zongertinib ("hot") drug substance and zongertinib, i.e. unlabelled ("cold") drug substance, and contained a radioactive dose of approximately 0.03 MBq.
  Interventions: Drug: zongertinib; Drug: zongertinib (C-14)

INTERVENTIONS:
Drug: zongertinib (C-14) — Oral solution
  Other Names: BI 1810631 (C-14), Hernexeos®
  Arms: Part A - zongertinib (C-14) (T1)
Drug: zongertinib — Film-coated tablet
  Other Names: BI 1810631, Hernexeos®
  Arms: Part B - zongertinib (T2), then zongertinib (C-14) (R)
Drug: zongertinib (C-14) — Solution for infusion
  Other Names: BI 1810631 (C-14), Hernexeos®
  Arms: Part B - zongertinib (T2), then zongertinib (C-14) (R)

SUMMARY:
Part A - the primary objective is to assess the mass balance and total recovery of [14C]-radioactivity in urine and faeces after oral single dose administration of BI 1810631 (C-14) (test treatment T1) in healthy male subjects.

Part A - the secondary objective is to assess concentrations of BI 1810631 and [14C]-radioactivity in plasma.

Part B - the primary objective is to investigate the absolute bioavailability of BI 1810631 administered as film-coated tablet (test treatment T2, not radio-labelled) compared with BI 1810631 (C-14) (reference treatment R) administered as intravenous microtracer.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
2. Age of 18 to 55 years (inclusive)
3. Body mass index (BMI) of 18.0 to 30.0 kg/m2 (inclusive)
4. Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial

Exclusion Criteria:

1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 145 millimetre of mercury (mmHg), diastolic blood pressure outside the range of 45 to 90 mmHg, or pulse rate outside the range of 40 to 100 beats per minute (bpm)
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
6. Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
7. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
8. History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- ICON, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Grempler R, Joseph D, Gan G, Auclair AM, Tiessen RG, Maw HH, Laux R, Wind S, Roessner PM, Sadrolhefazi B, Muller F, Minich D. Absorption, Metabolism, Distribution and Excretion (ADME) and Absolute Bioavailability Assessment of Zongertinib in Healthy Male Volunteers. Clin Drug Investig. 2025 Dec 5. doi: 10.1007/s40261-025-01509-9. Online ahead of print. PMID 41348300
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part A was an open-label, single-arm, single-dose part to investigate the pharmacokinetics of zongertinib and [14C]-radioactivity following one oral dose of zongertinib (C-14) containing a radioactive dose of approximately 3.7 Megabecquerel (MBq).
  Part B was an open-label, single-arm, single-period part to compare zongertinib administered orally to the intravenous infusion 2 hours later of zongertinib (C-14) solution (radioactive dose was approximately 0.03 MBq).
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | Part A - Zongertinib (C-14) (T1) | Part B - Zongertinib (T2), Then Zongertinib (C-14) (R)
Started | 8 | 7
Treated | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS) included all subjects who were treated with at least one dose of trial drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A - Zongertinib (C-14) (T1) | Part B - Zongertinib (T2), Then Zongertinib (C-14) (R) | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.8 (8.9) | 29.3 (8.5) | 28.5 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 7 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 7 | 14
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part A - Fraction Excreted in Urine and Faeces as Percentage of the Administered Dose Over the Time Interval From 0 to the Last Quantifiable Time Point (fe0-tz)
Description: Mass balance and total recovery of [14C]-radioactivity: fraction excreted in urine and faeces given as percentage of the administered oral dose of zongertinib (assessed by [14C]zongertinib-equivalent[EQ]) over the time interval from 0 to the last quantifiable time point (feurine, 0-tz; fefaeces, 0-tz) is reported.
  Timeframe (continued): after 336 h, if warranted, 24 h collections were to be performed every 7 days on days 21, 28, 35, and 42. Sampling was stopped when the release criteria for radioactivity recovery were met (earliest stopping on Day 15).
Time Frame: Within 18 h (urine) or 48 h (faeces) before drug intake; at 0-4, 4-8, 8-12, 12-24 (urine); and at 24 h sampling intervals until 336 h after drug intake (both). Both: after 336 h, every 7 days, up to day 42. Continues in description.
Population: Pharmacokinetic (PK) parameter analysis set (PKS) restricted to Part A included all part A subjects in the TS who provided at least one PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of the administered dose
Arm/Group | Part A - Zongertinib (C-14) (T1)
Number analyzed (Participants) | 8
Percentage of the administered dose
  feurine, 0-tz | 1.30 (16.8)
  fefaeces, 0-tz | 92.5 (3.66)
  feurine + fefaeces, 0-tz | 93.8 (3.62)

2. Primary Outcome: Part B - Dose-normalised Area Under the Concentration-time Curve in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞,Norm)
Description: The dose-normalised area under the concentration-time curve in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞,norm) after oral administration of zongertinib, and after intravenous administration of [14C]zongertinib, is reported.
  Geometric least square mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model, which included the effect 'subjects' as a random effect and 'treatment' as a fixed effect. These quantities were then back-transformed to the original scale.
Time Frame: Within 3 h prior and 0.5, 1, 1.5, 2, 2.5, 3, [zongertinib], 2, 2.08, 2.16, 2.25, 2.5, 2.75, 3, 3.5 [[14C]zongertinib], 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, and 168 h [zongertinib and [14C]zongertinib] after first drug administration.
Population: PKS restricted to Part B included all part B subjects in the TS who provided at least one PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Least Squares Mean (Standard Error); unit: hour*millimole/Liter/kilogram
Arm/Group | Part B - Zongertinib (T2), Then Zongertinib (C-14) (R)
Number analyzed (Participants) | 7
hour*millimole/Liter/kilogram
  zongertinib | 223.39 (NA) — Adjusted geometric standard error = 1.07
  [14C]zongertinib | 293.26 (NA) — Adjusted geometric standard error = 1.07
Statistical Analysis 1: Comparison: Part B - Zongertinib (T2), Then Zongertinib (C-14) (R); Ratio of adjusted geometric means was calculated using an ANOVA model on the logarithmic scale. The PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model, which included the effect 'subjects' as a random effect and 'treatment' as a fixed effect. These quantities were then back-transformed to the original scale; Test type: Other; Ratio of adjusted geometric means [%] = 76.18, 90% CI 2-sided [70.21 to 82.65] — Ratio [%] = (adjusted geometric mean zongertinib / adjusted geometric mean [14C]zongertinib)*100. Intra-individual geometric coefficient of variation (gCV) [%] = 7.9

3. Secondary Outcome: Part A - Maximum Measured Concentration of Zongertinib in Plasma (Cmax)
Description: Maximum measured concentration of zongertinib in plasma (Cmax) is reported.
Time Frame: Within 3 h prior and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 168, 216, 264, 336 h after drug administration.
Population: PKS restricted to Part A included all part A subjects in the TS who provided at least one PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/Liter
Arm/Group | Part A - Zongertinib (C-14) (T1)
Number analyzed (Participants) | 8
nanomole/Liter | 1160 (17.2)

4. Secondary Outcome: Part A - Maximum Measured Concentration of [14C]-Radioactivity (Assessed by [14C]Zongertinib-EQ) in Plasma (Cmax)
Description: Maximum measured concentration of [14C]-radioactivity (assessed by [14C]zongertinib-EQ) in plasma (Cmax) is reported.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/Liter
Arm/Group | Part A - Zongertinib (C-14) (T1)
Number analyzed (Participants) | 8
nanomole/Liter | 1450 (18.8)

5. Secondary Outcome: Part A - Area Under the Concentration-time Curve of Zongertinib in Plasma Over the Time Interval From 0 to the Last Quantifiable Time Point (AUC0-tz)
Description: Area under the concentration-time curve of zongertinib in plasma over the time interval from 0 to the last quantifiable time point (AUC0-tz) is reported.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanomole/Liter
Arm/Group | Part A - Zongertinib (C-14) (T1)
Number analyzed (Participants) | 8
hour*nanomole/Liter | 14100 (14.0)

6. Secondary Outcome: Part A - Area Under the Concentration-time Curve of [14C]-Radioactivity (Assessed by [14C]Zongertinib-EQ) in Plasma Over the Time Interval From 0 to the Last Quantifiable Time Point (AUC0-tz)
Description: Area under the concentration-time curve of [14C]-radioactivity (assessed by [14C]zongertinib-EQ) in plasma over the time interval from 0 to the last quantifiable time point (AUC0-tz) is reported.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanomole/Liter
Arm/Group | Part A - Zongertinib (C-14) (T1)
Number analyzed (Participants) | 8
hour*nanomole/Liter | 23700 (17.3)

7. Secondary Outcome: Part B - Dose-normalised Maximum Measured Concentration in Plasma (Cmax,Norm)
Description: The dose-normalised maximum measured concentration in plasma (Cmax,norm) after oral administration of zongertinib, and after intravenous administration of [14C]zongertinib, is reported.
  Geometric least square mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an ANOVA model on the logarithmic scale. The PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model, which included the effect 'subjects' as a random effect and 'treatment' as a fixed effect. These quantities were then back-transformed to the original scale.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Least Squares Mean (Standard Error); unit: picomole/Liter/microgram
Arm/Group | Part B - Zongertinib (T2), Then Zongertinib (C-14) (R)
Number analyzed (Participants) | 7
picomole/Liter/microgram
  zongertinib | 16.57 (NA) — Adjusted geometric standard error = 1.10
  [14C]zongertinib | 63.50 (NA) — Adjusted geometric standard error = 1.10
Statistical Analysis 1: Comparison: Part B - Zongertinib (T2), Then Zongertinib (C-14) (R); [analysis description as in outcome 2, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 26.10, 90% CI 2-sided [22.12 to 30.79] — Ratio [%] = (adjusted geometric mean zongertinib / adjusted geometric mean [14C]zongertinib)*100. Intra-individual geometric coefficient of variation (gCV) [%] = 16.0

8. Secondary Outcome: Part B - Dose-normalised Area Under the Concentration-time Curve in Plasma Over the Time Interval From 0 to the Last Quantifiable Time Point (AUC0-tz,Norm)
Description: The dose-normalised area under the concentration-time curve in plasma over the time interval from 0 to the last quantifiable time point (AUC0-tz,norm) after oral administration of zongertinib, and after intravenous administration of [14C]zongertinib, is reported.
  Geometric least square mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an ANOVA model on the logarithmic scale. The PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model, which included the effect 'subjects' as a random effect and 'treatment' as a fixed effect. These quantities were then back-transformed to the original scale.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Least Squares Mean (Standard Error); unit: hour*millimole/Liter/kilogram
Arm/Group | Part B - Zongertinib (T2), Then Zongertinib (C-14) (R)
Number analyzed (Participants) | 7
hour*millimole/Liter/kilogram
  zongertinib | 219.72 (NA) — Adjusted geometric standard error = 1.07
  [14C]zongertinib | 285.38 (NA) — Adjusted geometric standard error = 1.07
Statistical Analysis 1: Comparison: Part B - Zongertinib (T2), Then Zongertinib (C-14) (R); [analysis description as in outcome 2, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 76.99, 90% CI 2-sided [70.92 to 83.59] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: From the time of drug administration (part A), or of first drug administration (part B), up to 14 days. All-cause mortality: from first drug administration until the end of trial, up to approximately 6 (part A) or 3 (part B) weeks.
Description: Treated set (TS) included all subjects who were treated with at least one dose of trial drug.
Arm/Group | Part A - Zongertinib (C-14) (T1) | Part B - Zongertinib (T2), Then Zongertinib (C-14) (R)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 7/8 | 2/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A - Zongertinib (C-14) (T1) (N=8) | Part B - Zongertinib (T2), Then Zongertinib (C-14) (R) (N=7)
Impetigo (Infections and infestations) | 4 | 0
Tonsillitis (Infections and infestations) | 2 | 0
Pharyngotonsillitis (Infections and infestations) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 0
Catheter site bruise (General disorders) | 0 | 1
Catheter site haematoma (General disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-04-21): https://cdn.clinicaltrials.gov/large-docs/91/NCT05879991/Prot_002.pdf
  • Statistical Analysis Plan (2023-11-15): https://cdn.clinicaltrials.gov/large-docs/91/NCT05879991/SAP_001.pdf